CLINICAL TRIAL: NCT02389062
Title: Noninvasive Markers of Gluten Ingestion in Celiac Disease Patients: Prospective, Randomized,Placebo Controlled, Double Blind Clinical Trial
Brief Title: Noninvasive Markers of Gluten Ingestion in Celiac Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Jeff GI, Professor, Chair, Division of Gastroenterology, Director, celiac disease center, Thomas Jefferson University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 14D.389
Record Dates: First submitted 2015-02-12; First posted 2015-03-17 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Adult Form of Celiac Disease
MeSH Terms: interventions — Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo controlled group (Experimental): This is a group of same number of subjects as in other arms, who will be given equivalent dose of placebo- cornstarch capsules i.e 5 capsules containing neutral substance- cornstarch(placebo) to be taken daily by mouth for a period of 12 weeks.
  Interventions: Other: Administration of gluten( food /wheat protein) capsules or placebo(cornstarch) capsules and tests for novel markers will be done at intervals.
- High dose gluten capsules (Experimental): This group of subjects will be given high dose i.e 2.5 g of gluten containing capsules, 5 capsules to be taken daily by mouth, for a period of 12 weeks.
  Interventions: Other: Administration of gluten( food /wheat protein) capsules or placebo(cornstarch) capsules and tests for novel markers will be done at intervals.
- Low dose gluten capsules (Experimental): This group of subjects will be given low dose i.e 0.5 g of gluten containing capsules, 5 capsules to be taken daily by mouth, for a period of 12 weeks.
  Interventions: Other: Administration of gluten( food /wheat protein) capsules or placebo(cornstarch) capsules and tests for novel markers will be done at intervals.

INTERVENTIONS:
Other: Administration of gluten( food /wheat protein) capsules or placebo(cornstarch) capsules and tests for novel markers will be done at intervals. — After administering the capsules for 16 weeks during study periods, patients's blood will be tested for novel markers- Intestinal fatty acid binding protein(I-FABP), stool for gluten intestinal peptide (GIP), urine for gluten intestinal peptide(GIP), patient estimated gluten intake(PEGI), celiac severity index(CSI), Celiac dietary adherence test(CDAT) by standard questionnaire provided during the visits. These tests will be done over a period of 16 weeks and at a follow up 3 months later.

SUMMARY:
This is a clinical trial to evaluate the sensitivity of noninvasive, novel markers of gluten ingestion in celiac disease patients who are following gluten free diet for at least a period of one year. These noninvasive markers may be helpful to monitor the silent intestinal damage, possibly resulting from the accidental consumption of gluten due to cross contamination of gluten free diet.

DETAILED DESCRIPTION:
The gold-standard for monitoring of dietary adherence is consultation with an expert dietitian, but this may be time-consuming for patients and local expertise may not be available. Intestinal biopsy is the only direct method to document mucosal healing and can be considered in all adults with celiac disease. Non-invasive assessment of compliance with a gluten free diet(GFD) can be achieved with monitoring of IgA antibodies to tissue transglutaminase (IgA-tTG) or deamidated gliadin peptides, as these markers improve with gluten elimination. However, intestinal mucosal damage is present in a significant number of patients who report compliance with a gluten free diet and have normalized serology, potentially due to dietary lapses or unrecognized contamination with gluten. Furthermore, serologic testing may be normal in patients with partial adherence. Patient reported surveys show promise for assessing gluten free diet adherence, but further studies are needed.

Intestinal fatty acid-binding protein (I-FABP), a small (15 kD) cytosolic protein found exclusively in the small bowel enterocytes, has been studied as a marker of intestinal epithelial damage in septic shock and mesenteric ischemia. More recently, elevated levels of intestinal fatty acid-binding protein( I-FABP) have been described as a marker of intestinal injury in both adults and children with celiac disease. Intestinal fatty acid binding protein, (I-FABP) levels have been shown to significantly correlate with the degree of villous atrophy and IgA antibody to tissue transglutaminase (IgA-tTG), as well as decrease upon treatment with a gluten free diet(GFD). Incomplete normalization of intestinal fatty acid binding protein(I-FABP) on a gluten free diet points to ongoing intestinal injury, even in the absence of circulating antibodies, thus suggesting its potential as a non-invasive marker for gluten free diet adherence and intestinal damage in celiac disease.

The measurement of gluten immunogenic peptides (GIP) in stool is a novel method to monitor gluten free diet compliance. Recently, a technique to detect gliadin 33-mer equivalent peptide epitopes (33EPs) in the stool of pediatric patients has been described. These peptides show significant resistance to digestion and were detected in healthy individuals after normal gluten-containing diet ingestion. Importantly, these peptides are not detected in patients on a gluten free diet, and there appears to be a correlation between the amount of gluten intake and the peptide levels. A similar test has been developed for gluten intestinal peptide(GIP) detection in urine, although there are currently no peer-reviewed studies examining this technique. Further research on the utility of stool and urine gluten intestinal peptide (GIP)for monitoring of gluten free diet (GFD) adherence is warranted.

Given the lack of a non-invasive and accurate measure of gluten intake in celiac disease (CD), the investigators will investigate the effect of gluten intake in celiac disease (CD) patients using a variety of markers. Patients who are symptom-free on a gluten free diet (GFD) will be exposed to various amounts of gluten. Factors that will be studied include the effect on patient estimated gluten intake, Celiac disease symptoms, IgA-tTG level,intestinal fatty acid binding protein( I-FABP) level, and both stool and urine gluten peptide levels.

ELIGIBILITY:
Inclusion Criteria:

* This study population will consist of patients with a prior diagnosis of celiac disease based on intestinal biopsy (Marsh score of 1-4) who report control of symptoms with adherence to gluten free diet(GFD) for at least one year and have a baseline IgA antibody to tissue transglutaminase(IgA-tTG) within the normal range.

Exclusion Criteria:

* Patients < 18 years of age
* Patients with refractory celiac disease (RFD), defined as persisting or recurring symptoms and mucosal villous atrophy, despite strict adherence to a gluten free diet (GFD) for >12 months and a negative IgA antibody to tissue transglutaminase (IgA-tTG)
* Patients with enteropathy-associated T-cell lymphoma
* Patients with IgA deficiency
* Patients with a diagnosis of inflammatory bowel disease, irritable bowel symptoms, or acute gastroenteritis
* Patients taking immunosuppressive medications
* Patients who are pregnant
* Patients who are breast feeding/lactating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-02-11 (Actual); Primary Completion 2016-02-11 (Actual); Study Completion 2017-02-11 (Actual)

PRIMARY OUTCOMES:
1) Change in the patient estimated gluten intake after administration of study pills using the Celiac Dietary Adherence Test (CDAT), to be assessed at the end of follow up week 12 | up to follow up week 12
Change in the Celiac disease symptoms, using the Celiac Symptom Index (CSI) after administration of study pills; to be assessed at the end of follow up week 12 | up to follow up week 12
  questionnaire
Change in IgA antibody to tissue transglutaminase (IgA-TTG) levels after administration of study pills, to be assessed at the end of follow up week 12. | up to follow up week 12
  lab
Change in Intestinal fatty acid binding protein (I-FABP) levels after administration of study pills, to be assessed at the end of follow up week 12. | up to follow up week 12
  lab
Change in stool gluten intestinal peptide (GIP) level after administration of study pills, to be assessed at the end of follow up week 12 | up to follow up week 12
  lab
Change in urine gluten intestinal peptide (GIP) level after administration of study pills,to be assessed at the end of follow up week 12 | up to follow up week 12
  lab
Change in patient estimated gluten intake(PEGI) after administration of study pills, using separate questionnaire, to be assessed at the end of follow up week 12 | up to follow up week 12
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J. DiMarino, MD, Principal Investigator — Thomas Jefferson University, Philadelphia, PA 19107
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Rubio-Tapia A, Hill ID, Kelly CP, Calderwood AH, Murray JA; American College of Gastroenterology. ACG clinical guidelines: diagnosis and management of celiac disease. Am J Gastroenterol. 2013 May;108(5):656-76; quiz 677. doi: 10.1038/ajg.2013.79. Epub 2013 Apr 23. PMID 23609613
- [Background] Murray JA, Watson T, Clearman B, Mitros F. Effect of a gluten-free diet on gastrointestinal symptoms in celiac disease. Am J Clin Nutr. 2004 Apr;79(4):669-73. doi: 10.1093/ajcn/79.4.669. PMID 15051613
- [Background] Lee SK, Lo W, Memeo L, Rotterdam H, Green PH. Duodenal histology in patients with celiac disease after treatment with a gluten-free diet. Gastrointest Endosc. 2003 Feb;57(2):187-91. doi: 10.1067/mge.2003.54. PMID 12556782
- [Background] Rubio-Tapia A, Rahim MW, See JA, Lahr BD, Wu TT, Murray JA. Mucosal recovery and mortality in adults with celiac disease after treatment with a gluten-free diet. Am J Gastroenterol. 2010 Jun;105(6):1412-20. doi: 10.1038/ajg.2010.10. Epub 2010 Feb 9. PMID 20145607
- [Background] Bai JC, Gonzalez D, Mautalen C, Mazure R, Pedreira S, Vazquez H, Smecuol E, Siccardi A, Cataldi M, Niveloni S, Boerr LA, Maurino E. Long-term effect of gluten restriction on bone mineral density of patients with coeliac disease. Aliment Pharmacol Ther. 1997 Feb;11(1):157-64. doi: 10.1046/j.1365-2036.1997.112283000.x. PMID 9042988
- [Background] Dickey W. Low serum vitamin B12 is common in coeliac disease and is not due to autoimmune gastritis. Eur J Gastroenterol Hepatol. 2002 Apr;14(4):425-7. doi: 10.1097/00042737-200204000-00016. PMID 11943958
- [Background] Halfdanarson TR, Kumar N, Hogan WJ, Murray JA. Copper deficiency in celiac disease. J Clin Gastroenterol. 2009 Feb;43(2):162-4. doi: 10.1097/MCG.0b013e3181354294. PMID 18496230
- [Background] Kotze LM. Gynecologic and obstetric findings related to nutritional status and adherence to a gluten-free diet in Brazilian patients with celiac disease. J Clin Gastroenterol. 2004 Aug;38(7):567-74. doi: 10.1097/01.mcg.0000131720.90598.6a. PMID 15232359
- [Background] Choi JM, Lebwohl B, Wang J, Lee SK, Murray JA, Sauer MV, Green PH. Increased prevalence of celiac disease in patients with unexplained infertility in the United States. J Reprod Med. 2011 May-Jun;56(5-6):199-203. PMID 21682114
- [Background] Khashan AS, Henriksen TB, Mortensen PB, McNamee R, McCarthy FP, Pedersen MG, Kenny LC. The impact of maternal celiac disease on birthweight and preterm birth: a Danish population-based cohort study. Hum Reprod. 2010 Feb;25(2):528-34. doi: 10.1093/humrep/dep409. Epub 2009 Nov 24. PMID 19939833
- [Background] Catassi C, Fabiani E, Iacono G, D'Agate C, Francavilla R, Biagi F, Volta U, Accomando S, Picarelli A, De Vitis I, Pianelli G, Gesuita R, Carle F, Mandolesi A, Bearzi I, Fasano A. A prospective, double-blind, placebo-controlled trial to establish a safe gluten threshold for patients with celiac disease. Am J Clin Nutr. 2007 Jan;85(1):160-6. doi: 10.1093/ajcn/85.1.160. PMID 17209192
- [Background] Haines ML, Anderson RP, Gibson PR. Systematic review: The evidence base for long-term management of coeliac disease. Aliment Pharmacol Ther. 2008 Nov 1;28(9):1042-66. doi: 10.1111/j.1365-2036.2008.03820.x. Epub 2008 Jul 30. PMID 18671779
- [Background] Nachman F, Sugai E, Vazquez H, Gonzalez A, Andrenacci P, Niveloni S, Mazure R, Smecuol E, Moreno ML, Hwang HJ, Sanchez MI, Maurino E, Bai JC. Serological tests for celiac disease as indicators of long-term compliance with the gluten-free diet. Eur J Gastroenterol Hepatol. 2011 Jun;23(6):473-80. doi: 10.1097/MEG.0b013e328346e0f1. PMID 21537123
- [Background] Lanzini A, Lanzarotto F, Villanacci V, Mora A, Bertolazzi S, Turini D, Carella G, Malagoli A, Ferrante G, Cesana BM, Ricci C. Complete recovery of intestinal mucosa occurs very rarely in adult coeliac patients despite adherence to gluten-free diet. Aliment Pharmacol Ther. 2009 Jun 15;29(12):1299-308. doi: 10.1111/j.1365-2036.2009.03992.x. Epub 2009 Mar 3. PMID 19302264
- [Background] Vahedi K, Mascart F, Mary JY, Laberenne JE, Bouhnik Y, Morin MC, Ocmant A, Velly C, Colombel JF, Matuchansky C. Reliability of antitransglutaminase antibodies as predictors of gluten-free diet compliance in adult celiac disease. Am J Gastroenterol. 2003 May;98(5):1079-87. doi: 10.1111/j.1572-0241.2003.07284.x. PMID 12809831
- [Background] Leffler DA, Edwards George JB, Dennis M, Cook EF, Schuppan D, Kelly CP. A prospective comparative study of five measures of gluten-free diet adherence in adults with coeliac disease. Aliment Pharmacol Ther. 2007 Nov 1;26(9):1227-35. doi: 10.1111/j.1365-2036.2007.03501.x. PMID 17944737
- [Background] Leffler DA, Dennis M, Edwards George JB, Jamma S, Magge S, Cook EF, Schuppan D, Kelly CP. A simple validated gluten-free diet adherence survey for adults with celiac disease. Clin Gastroenterol Hepatol. 2009 May;7(5):530-6, 536.e1-2. doi: 10.1016/j.cgh.2008.12.032. Epub 2009 Jan 11. PMID 19268725
- [Background] Derikx JP, Poeze M, van Bijnen AA, Buurman WA, Heineman E. Evidence for intestinal and liver epithelial cell injury in the early phase of sepsis. Shock. 2007 Nov;28(5):544-8. doi: 10.1097/shk.0b013e3180644e32. PMID 17607153
- [Background] Lieberman JM, Sacchettini J, Marks C, Marks WH. Human intestinal fatty acid binding protein: report of an assay with studies in normal volunteers and intestinal ischemia. Surgery. 1997 Mar;121(3):335-42. doi: 10.1016/s0039-6060(97)90363-9. PMID 9068676
- [Background] Kanda T, Fujii H, Tani T, Murakami H, Suda T, Sakai Y, Ono T, Hatakeyama K. Intestinal fatty acid-binding protein is a useful diagnostic marker for mesenteric infarction in humans. Gastroenterology. 1996 Feb;110(2):339-43. doi: 10.1053/gast.1996.v110.pm8566578.
- [Background] Kanda T, Tsukahara A, Ueki K, Sakai Y, Tani T, Nishimura A, Yamazaki T, Tamiya Y, Tada T, Hirota M, Hasegawa J, Funaoka H, Fujii H, Hatakeyama K. Diagnosis of ischemic small bowel disease by measurement of serum intestinal fatty acid-binding protein in patients with acute abdomen: a multicenter, observer-blinded validation study. J Gastroenterol. 2011 Apr;46(4):492-500. doi: 10.1007/s00535-011-0373-2. Epub 2011 Feb 5. PMID 21298292
- [Background] Derikx JP, Vreugdenhil AC, Van den Neucker AM, Grootjans J, van Bijnen AA, Damoiseaux JG, van Heurn LW, Heineman E, Buurman WA. A pilot study on the noninvasive evaluation of intestinal damage in celiac disease using I-FABP and L-FABP. J Clin Gastroenterol. 2009 Sep;43(8):727-33. doi: 10.1097/MCG.0b013e31819194b0. PMID 19359998
- [Background] Vreugdenhil AC, Wolters VM, Adriaanse MP, Van den Neucker AM, van Bijnen AA, Houwen R, Buurman WA. Additional value of serum I-FABP levels for evaluating celiac disease activity in children. Scand J Gastroenterol. 2011 Dec;46(12):1435-41. doi: 10.3109/00365521.2011.627447. Epub 2011 Oct 27. PMID 22029621
- [Background] Adriaanse MP, Tack GJ, Passos VL, Damoiseaux JG, Schreurs MW, van Wijck K, Riedl RG, Masclee AA, Buurman WA, Mulder CJ, Vreugdenhil AC. Serum I-FABP as marker for enterocyte damage in coeliac disease and its relation to villous atrophy and circulating autoantibodies. Aliment Pharmacol Ther. 2013 Feb;37(4):482-90. doi: 10.1111/apt.12194. Epub 2013 Jan 7. PMID 23289539
- [Background] Rodriguez-Herrera A, Comino I, Real A, et al, Monitoring of gluten-free diet compliance in pediatric patients by fecal check; (Abstract #F613). Presented at the 15th International Celiac Disease Symposium. September, 2013. Chicago.
- [Background] Comino I, Real A, Vivas S, Siglez MA, Caminero A, Nistal E, Casqueiro J, Rodriguez-Herrera A, Cebolla A, Sousa C. Monitoring of gluten-free diet compliance in celiac patients by assessment of gliadin 33-mer equivalent epitopes in feces. Am J Clin Nutr. 2012 Mar;95(3):670-7. doi: 10.3945/ajcn.111.026708. Epub 2012 Jan 18. PMID 22258271
- [Background] Leffler DA, Dennis M, Edwards George J, Jamma S, Cook EF, Schuppan D, Kelly CP. A validated disease-specific symptom index for adults with celiac disease. Clin Gastroenterol Hepatol. 2009 Dec;7(12):1328-34, 1334.e1-3. doi: 10.1016/j.cgh.2009.07.031. Epub 2009 Aug 7. PMID 19665584
- [Result] Fasano A, Catassi C. Clinical practice. Celiac disease. N Engl J Med. 2012 Dec 20;367(25):2419-26. doi: 10.1056/NEJMcp1113994. No abstract available. PMID 23252527